CLINICAL TRIAL: NCT00349739
Title: Clinical Treatment of Patients With Age-Related Macular Degeneration With Anecortave Acetate Sterile Suspension
Brief Title: Treatment of Patients With Age-Related Macular Degeneration With Anecortave Acetate
Status: No longer available | Type: Expanded Access
Sponsor: University of Iowa (Other)
Responsible Party: Edwin M. Stone, MD, PHD, Professor, Principal investigator, University of Iowa
Other Study IDs: UIOWA200101096; AL-3789
Record Dates: First submitted 2006-07-06; First posted 2006-07-10 (Estimated); Last update posted 2010-01-15 (Estimated); Status verified 2010-01

CONDITIONS: Macular Degeneration
Keywords: age related macular degeneration
MeSH Terms: conditions — Macular Degeneration | interventions — anecortave acetate

INTERVENTIONS:
Drug: Anecortave Acetate — Dosage: 0.5ml of 30mg/ml(15 mg) or 60mg/ml(30mg) Duration of action: 159-180 days
  Other Names: Retaane

SUMMARY:
The purpose of this study is to evaluate whether anecortave acetate can slow or stop the progression of age-related macular degeneration in patients who do not qualify for other studies and have no other treatment options.

DETAILED DESCRIPTION:
Choroidal neovascularization (CNV), a complication of age-related macular degeneration (AMD), is the most common cause of profound visual loss in the United States. Laser photocoagulation has been shown to retard visual loss, however only about 20% of patients with CNV are eligible for laser treatment.

Conventional laser photocoagulation of CNV requires laser intensities adequate to coagulate proteins in the target tissue. Due to the proximity of CNV to the center of vision (fovea), the intensity of laser irradiation necessary, and the heat conduction in the ocular tissues, collateral tissue damage often results which further compromises vision. Recently, a new class of compounds (angiostatic steroids) have been found to inhibit the formation of new blood vessels (i.e. neovascularization) in the eye. One new angiostatic steroid, anecortave acetate (AL-3789), may represent a breakthrough in the therapy of ocular neovascular diseases such as AMD and diabetic retinopathy. Anecortave acetate suppresses the formation of new blood vessels in a variety of models of neovascularization. Unlike some of the angiostatic steroids, anecortave acetate appears to be lacking in the pharmacological activities typical of the steroid family (i.e. glucocorticoid, anti-inflammatory, cardiovascular, neurologic, diuretic, etc.) Additionally, anecortave acetate has been shown to arrest lipopolysaccharide (LPS) and basic fibroblast growth factors (bFGH) induced corneal neovascularization, to attenuate oxygen-induced retinopathy and to inhibit the growth of a highly vascularized intraocular tumor.

The purpose of this study is to treat a small number of patients who would not normally qualify for the other anecortave acetate studies. These patients who are not eligible for the other anecortave acetate studies have no other treatment options and will likely experience a poor visual outcome as a result of their AMD. These patients are excluded from other studies because of "occult" neovascularization and visual acuity worse than 20/40. Sub-Tenon's injection of either 15 mg or 30 mg of anecortave acetate will be administered at the University of Iowa. The patients will be followed for a minimum of 24 months.

ELIGIBILITY:
Inclusion Criteria:

* Choroidal neovascularization, mostly occult
* Visual acuity > 20/40 in study eye

Exclusion Criteria:

* Allergy to fluorescein dye
* Inability to stop warfarin prior to treatment
* Pregnancy
* Other serious ocular diseases or conditions

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2003-01; Study Completion 2008-08 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Edwin M Stone, MD, PhD, Principal Investigator — University of Iowa; Stephen R. Russell, MD, Study Director — University of Iowa
Locations (1):
- University of Iowa Hospitals and Clinics, Ophthalmology, Iowa City, Iowa, United States

REFERENCES:
- See also: Laboratory Website — http://cmd.ophth.uiowa.edu/